CLINICAL TRIAL: NCT03072563
Title: The Use of the Cerebro-placental Ratio to Predict Adverse Outcomes in Pregnancies Complicated by Gestational Diabetes
Brief Title: The Use of the CPR to Predict Adverse Outcomes in GDM Pregnancies
Acronym: CPR GDM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Unity Health Toronto (Other)
Responsible Party: Sponsor
Other Study IDs: 16-382
Record Dates: First submitted 2017-03-02; First posted 2017-03-07 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Gestational Diabetes
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The cerebro-placental ratio (CPR) is a tool for assessment of fetal wellbeing in the management of the growth restricted fetus. CPR is the ratio of the fetal middle cerebral artery pulsatility index (PI) to the umbilical artery PI. In Gestational Diabetes (GDM), the common finding is of accelerated and asymmetric fetal growth. Pregnancies complicated by GDM have an increased risk of certain complications such as preeclampsia, intrauterine demise, CS due to fetal distress. These complications have a well known association with fetal growth restriction leading to the hypothesis that there exists a subset of diabetic fetuses that exhibit a growth restriction phenotype despite not being small for gestational age (<10%).The objective of this study is to examine whether the CPR can identify GDM fetuses that are not growth restricted but are at increased risk of certain adverse neonatal outcomes. Women with singleton pregnancies and a diagnosis of GDM at 24 weeks of gestation and beyond will be included. Exclusion criteria are Pre-gestational diabetes, hypertensive disease of pregnancy at time of recruitment, fetus with a known major anomaly, fetal EFW < 10%(IUGR). Women who consent to the study will have a blinded Doppler assessment of CPR. Clinicians will be blinded to these Doppler measurements (unless they are indicated clinically for another reason (suspected fetal anemia or IUGR development- and the results will be unblinded and reported to the clinicians). Obstetric and neonatal outcomes will be collected prospctively via the local BORN database and the patient chart. Local BORN is needed for the registered outcomes. Newborns will be divided post-hoc into two groups: A) last CPR <10% B) Last CPR > 10%. The primary outcome will be a composite outcome consisting of one or more of the following: Caesarean section due to suspected fetal distress, 5 minute Apgar <7, Cord arterial PH < 7, HIE, NICU admission >24 hours.

ELIGIBILITY:
Inclusion Criteria:

* All women over the age of 18 years old with singleton pregnancies and a diagnosis of GDM at 24 weeks of gestation and beyond.

Exclusion Criteria:

* Pre-gestational diabetes, Hypertensive disease of pregnancy at time of recruitment, fetus with a known major anomaly, fetal EFW < 10% or suspected fetal anemia (and thus requiring a clinically indicated CPR measurement) poor grasp of english

Ages: 18 Years to 45 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes — pregnant females
Study Population: Pregnant women diagnosed with gestational diabetes.
Sampling Method: Non-Probability Sample
Enrollment: 207 (Estimated)
Dates: Start 2017-03-07 (Actual); Primary Completion 2021-03-07 (Estimated); Study Completion 2021-03-07 (Estimated)

PRIMARY OUTCOMES:
Composite outcome | 24 weeks gestation to delivery
  Caesarean section due to suspected fetal distress, 5 minute Apgar <7, Cord arterial PH < 7, HIE, NICU admission >24 hours

CONTACTS AND LOCATIONS:
Locations (1):
- St. Michael's Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No